CLINICAL TRIAL: NCT00655941
Title: Influence of Weight Loss or Exercise on CARtilage in Obese Knee Osteoarthritis Patients: a Randomized Controlled Trial (CAROT).
Brief Title: Influence of Weight Loss or Exercise on Cartilage in Obese Knee Osteoarthritis Patients
Acronym: CAROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henning Bliddal (Other)
Collaborators: Velux Fonden (Other); Oak Foundation (Other); The Danish Rheumatism Association (Other); Cambridge Weight Plan Limited (Industry)
Responsible Party: Sponsor-Investigator, Henning Bliddal, professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-B-2007-088
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Osteoarthritis, Knee; Obesity
Keywords: Osteoarthritis; Obesity; Weight loss; Dietary instruction; Exercise; Attention
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity; Osteoarthritis; Weight Loss; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Dietary instruction (low-energy diet. This is given by instructions in groups of 8
  Interventions: Behavioral: Dietary instruction
- 2 (Active Comparator): Exercise
  Interventions: Other: Exercise
- 3 (No Intervention): Control

INTERVENTIONS:
Behavioral: Dietary instruction — Weekly instruction by dieticians
  Other Names: The Cambridge Programme
  Arms: 1
Other: Exercise — Supervised exercise in groups
  Arms: 2

SUMMARY:
Obesity and osteoarthritis (OA) co-exist in an increasing part of the population.

The two diseases intertwine in several ways. The evolution in the population shows a tendency towards deterioration of both by increasing general age and weight. The two diseases share pathogenetic features and the development of one disease increases the risk of the other and may be the onset of a vicious circle.

There is a link between treatments of these two diseases as well. There is now solid (gold) evidence that by treating effectively the obesity of patients with co-occurring OA, the functional status is dramatically ameliorated; the short-term results are equal to that of a joint replacement. The long-term efficacy of a weight loss remains to be shown. OA is definitely one of many diseases in which obesity must be taken seriously into account when planning a correct treatment of patients. This trial has two phases, the first (16 weeks) consisting of a dietary intervention with low-energy diet and the second (52 weeks) a randomized, three group (each n>50 patients) controlled study of maintenance of weight loss by either continuing dietary instruction, exercise, or a control group. The hypothesis is that maintenance of an initially induced weight loss is dependent on attention rather than any specific therapy.

DETAILED DESCRIPTION:
Any patient with osteoarthritis (OA)of the knee and concomitant obesity will be considered for participation. Eligible for this study will be patients with radiographical knee OA. Exclusion criteria are recent or planned knee operations, alloplasties in both knees, ongoing or planned alternative interventions against obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI >=30
* Radiographical knee OA
* Age >=50
* Spoken Danish
* Motivated for weight loss

Exclusion Criteria:

* Bilateral Alloplasty of the knees
* Ongoing or planned surgery
* Ongoing or planned alternative weight loss programme
* Intellectual disability

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Pain | 16 weeks, 68 weeks
OMERACT-OARSI response criterion | 16 weeks, 68 weeks

SECONDARY OUTCOMES:
Weight change | 8 weeks, 16 weeks, 68 weeks
Gait analysis | 16 weeks, 68 weeks
MRI | 16 weeks, 68 weeks
Ultrasound | 16 weeks, 68 weeks
Collagen markers | 16 weeks, 68 weeks
Metabolic syndrome | 8 weeks, 16 weeks, 68 weeks
KOOS | 16 weeks, 68 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, Professor,MD, Study Director — The Parker Institute, Frederiksberg Hospital, Denmark
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Frederiksberg, Frederiksberg, Denmark

REFERENCES:
- [Background] Christensen R, Bartels EM, Astrup A, Bliddal H. Effect of weight reduction in obese patients diagnosed with knee osteoarthritis: a systematic review and meta-analysis. Ann Rheum Dis. 2007 Apr;66(4):433-9. doi: 10.1136/ard.2006.065904. Epub 2007 Jan 4. PMID 17204567
- [Background] Bliddal H, Christensen R. The management of osteoarthritis in the obese patient: practical considerations and guidelines for therapy. Obes Rev. 2006 Nov;7(4):323-31. doi: 10.1111/j.1467-789X.2006.00252.x. PMID 17038126
- [Background] Christensen R, Astrup A, Bliddal H. Weight loss: the treatment of choice for knee osteoarthritis? A randomized trial. Osteoarthritis Cartilage. 2005 Jan;13(1):20-7. doi: 10.1016/j.joca.2004.10.008. PMID 15639633
- [Background] Roddy E, Zhang W, Doherty M. Aerobic walking or strengthening exercise for osteoarthritis of the knee? A systematic review. Ann Rheum Dis. 2005 Apr;64(4):544-8. doi: 10.1136/ard.2004.028746. PMID 15769914
- [Derived] Bartels EM, Henrotin Y, Bliddal H, Centonze P, Henriksen M. Relationship between weight loss in obese knee osteoarthritis patients and serum biomarkers of cartilage breakdown: secondary analyses of a randomised trial. Osteoarthritis Cartilage. 2017 Oct;25(10):1641-1646. doi: 10.1016/j.joca.2017.06.009. Epub 2017 Jul 6. PMID 28689920
- [Derived] Christensen R, Henriksen M, Leeds AR, Gudbergsen H, Christensen P, Sorensen TJ, Bartels EM, Riecke BF, Aaboe J, Frederiksen R, Boesen M, Lohmander LS, Astrup A, Bliddal H. Effect of weight maintenance on symptoms of knee osteoarthritis in obese patients: a twelve-month randomized controlled trial. Arthritis Care Res (Hoboken). 2015 May;67(5):640-50. doi: 10.1002/acr.22504. PMID 25370359
- [Derived] Bartels EM, Christensen R, Christensen P, Henriksen M, Bennett A, Gudbergsen H, Boesen M, Bliddal H. Effect of a 16 weeks weight loss program on osteoarthritis biomarkers in obese patients with knee osteoarthritis: a prospective cohort study. Osteoarthritis Cartilage. 2014 Nov;22(11):1817-25. doi: 10.1016/j.joca.2014.07.027. Epub 2014 Aug 12. PMID 25106676
- [Derived] Henriksen M, Christensen R, Hunter DJ, Gudbergsen H, Boesen M, Lohmander LS, Bliddal H. Structural changes in the knee during weight loss maintenance after a significant weight loss in obese patients with osteoarthritis: a report of secondary outcome analyses from a randomized controlled trial. Osteoarthritis Cartilage. 2014 May;22(5):639-46. doi: 10.1016/j.joca.2014.03.003. Epub 2014 Mar 15. PMID 24636948
- [Derived] Henriksen M, Hunter DJ, Dam EB, Messier SP, Andriacchi TP, Lohmander LS, Aaboe J, Boesen M, Gudbergsen H, Bliddal H, Christensen R. Is increased joint loading detrimental to obese patients with knee osteoarthritis? A secondary data analysis from a randomized trial. Osteoarthritis Cartilage. 2013 Dec;21(12):1865-75. doi: 10.1016/j.joca.2013.10.003. Epub 2013 Oct 14. PMID 24135273
- [Derived] Gudbergsen H, Boesen M, Christensen R, Bartels EM, Henriksen M, Danneskiold-Samsoe B, Bliddal H. Changes in bone marrow lesions in response to weight-loss in obese knee osteoarthritis patients: a prospective cohort study. BMC Musculoskelet Disord. 2013 Mar 22;14:106. doi: 10.1186/1471-2474-14-106. PMID 23522337
- [Derived] Gudbergsen H. MRI in knee osteoarthritis. Application in diet intervention. Dan Med J. 2013 Mar;60(3):B4594. PMID 23484617
- [Derived] Gudbergsen H, Lohmander LS, Jones G, Christensen R, Bartels EM, Danneskiold-Samsoe B, Bliddal H, Boesen M. Correlations between radiographic assessments and MRI features of knee osteoarthritis--a cross-sectional study. Osteoarthritis Cartilage. 2013 Apr;21(4):535-43. doi: 10.1016/j.joca.2012.12.010. Epub 2012 Dec 26. PMID 23274104
- [Derived] Christensen P, Bartels EM, Riecke BF, Bliddal H, Leeds AR, Astrup A, Winther K, Christensen R. Improved nutritional status and bone health after diet-induced weight loss in sedentary osteoarthritis patients: a prospective cohort study. Eur J Clin Nutr. 2012 Apr;66(4):504-9. doi: 10.1038/ejcn.2011.201. Epub 2011 Dec 21. PMID 22190136
- [Derived] Henriksen M, Christensen R, Danneskiold-Samsoe B, Bliddal H. Changes in lower extremity muscle mass and muscle strength after weight loss in obese patients with knee osteoarthritis: a prospective cohort study. Arthritis Rheum. 2012 Feb;64(2):438-42. doi: 10.1002/art.33394. PMID 22161649
- [Derived] Gudbergsen H, Bartels EM, Krusager P, Waehrens EE, Christensen R, Danneskiold-Samsoe B, Bliddal H. Test-retest of computerized health status questionnaires frequently used in the monitoring of knee osteoarthritis: a randomized crossover trial. BMC Musculoskelet Disord. 2011 Aug 18;12:190. doi: 10.1186/1471-2474-12-190. PMID 21851618
- [Derived] Riecke BF, Christensen R, Christensen P, Leeds AR, Boesen M, Lohmander LS, Astrup A, Bliddal H. Comparing two low-energy diets for the treatment of knee osteoarthritis symptoms in obese patients: a pragmatic randomized clinical trial. Osteoarthritis Cartilage. 2010 Jun;18(6):746-54. doi: 10.1016/j.joca.2010.02.012. Epub 2010 Feb 17. PMID 20206314